CLINICAL TRIAL: NCT01538927
Title: Evaluation of Early Wound Healing Following Use of Fibrin Sealant (FS) in Periodontal Surgery. A Controlled Randomized Clinical Trial.
Brief Title: Effect of Fibrin Sealant on Early Wound Healing
Acronym: FS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chhattisgarh Dental College and Research Institute (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Dr Shaju Jacob P, Professor, Chhattisgarh Dental College and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDC0212-FS; CTRI/2012/05/002628 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2012-02-10; First posted 2012-02-24 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Periodontitis
Keywords: fibrin sealant; tissue adhesive; wound healing; interleukin 1 beta; interleukin 8
MeSH Terms: conditions — Periodontitis | interventions — Fibrin Tissue Adhesive; Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrin Sealant (Experimental): One quadrant surgically elevated will be closed with fibrin sealant
  Interventions: Drug: Fibrin Sealant
- Suture (Placebo Comparator): The surgically elevated flap is closed with non resorbable sutures.
  Interventions: Drug: Suture

INTERVENTIONS:
Drug: Fibrin Sealant — Fibrin Sealant 4ml (Baxter Tisseel)
  Other Names: TISSEEL™ Kit, Two component Fibrin Sealant, Steam - treated
  Arms: Fibrin Sealant
Drug: Suture — Black silk 000
  Other Names: Ethicon
  Arms: Suture

SUMMARY:
The aim of this randomized controlled clinical trial is to compare wound healing after the use of fibrin sealant and sutures for gum surgeries. 15 patients requiring gum surgery for their periodontal (gum)problems are selected and invited. Two regions will be operated in a selected patient. One region will receive fibrin sealant (test site) and the other region will get sutures (control site). Wound healing will be assessed by evaluating inflammatory markers, Interleukin 1beta and interleukin 8, from a non invasively collected gum fluid.

Hypothesis. Fibrin sealant use will result in less inflammation seen through reduced levels of interleukin (1beta and 8) compared to use of sutures.

ELIGIBILITY:
Inclusion Criteria:

1. A subject has to be between the ages of 18 and 60 years.
2. Severe Periodontitis: Presence of a jaw with each quadrant having atleast 4 teeth with a probing depth of ≥ 6mm and is indicated for periodontal flap surgery.
3. Compliance: Only patients with optimal compliance, as assessed during the cause-related phase of therapy, are selected.
4. Good oral hygiene: Full-mouth plaque score (FMPS) < 25%.
5. Low levels of residual infection: Full-mouth bleeding score (FMBS) < 25%.
6. Endodontic status: Teeth had to be vital or properly treated with root canal therapy

Exclusion Criteria:

1. History of any systemic disease such as diabetes mellitus, osteoporosis, unstable or life-threatening conditions, bleeding disorder, undergoing antibiotic or other antimicrobial therapy.
2. Current or former smokers.
3. Had undergone periodontal therapy in the past 6 months, or exhibit poor plaque control after phase I therapy.
4. Mobility of selected teeth.
5. Pregnant or lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Concentration of cytokines. | 7 days
  Assess the concentration of Interleukin 1beta and Interleukin 8 in GCF of test and control sites after 7 days.

SECONDARY OUTCOMES:
Clinical inflammation | 7, 14 and 21 days
  Gingival inflammation will be assessed at a clinical level.

CONTACTS AND LOCATIONS:
Overall Officials: Shaju P Jacob, MDS, Principal Investigator — Chhattisgarh Dental College and Research Institute
Locations (1):
- Chhattisgarh Dental College and Research Institute, Rāj-Nāndgaon, Chhattisgarh, India